CLINICAL TRIAL: NCT04736342
Title: Patients Acceptance Towards Elective Induction of Labor at 39th Week of Gestation (PALI)
Brief Title: Patients Acceptance Towards Elective Labor in Induction (PALI)
Acronym: PALI
Status: Completed | Type: Observational
Sponsor: Hanoi Obstetrics and Gynecology Hospital (Other)
Collaborators: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PSHN.0002.2021
Record Dates: First submitted 2021-01-22; First posted 2021-02-03 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Patient Acceptance of Health Care
Keywords: Patients Acceptance; Induction of Labor; PALI
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PALI questionaire — Survey comprised of a series of multiple choice questions

SUMMARY:
To assess patients' preference, understanding regarding elective IOL and factors contribute to decision making process towards elective IOL at 39th week of gestation.

DETAILED DESCRIPTION:
A normal pregnancy lasts between 37+0 to 41+6 weeks. Estimated date of delivery is set exactly at 40+0 weeks of gestation. Base on this estimation, professional society's guidelines have recommended to start inducing the labor from 41+0 to 41+6 weeks after the last menstrual period. Clinical practice during the last few decades has been moving towards this trend and postponing labor induction.

But is 40 weeks' gestational age the optimal endpoint of human pregnancy? Recent studies, however, showed different results where many of them support induction of labor at 39 weeks. A large cohort retrospective study which included information from merely 5.4 million non-anomalous live births in the United States from 2012 to 2016, though only modestly, the authors have been able to conclude that the rates of composite neonatal and maternal adverse outcomes increase from 39 through 41 weeks of gestation among low-risk parous women. Stratifying by parity, it seemed that the trend is also similar among all low-risk women no matter which parities they are in. When it comes to nulliparous women, results from a large prospective randomized control trial (the ARRIVE trial) show that induction of labor at 39 weeks in low-risk nulliparous women did not lead to significant lower frequency of a composite adverse perinatal outcome but it did result in a significant lower rate of cesarean delivery. More recently, in a review sponsored by the Cochrane library on induction of labor beyond 37 weeks' gestation has found that there is a clear reduction in perinatal death with a policy of labor induction at or beyond 37 weeks compared with expectant management, though absolute rates are small (0.4 versus 3 deaths per 1000). There were also lower caesarean rates without increasing rates of operative vaginal births and there were fewer Neonatal Intensive Care Unit admissions with a policy of induction. Base on these evidence, the American College of Obstetricians and Gynecologists has suggested "it's time to induce of labor at 39th week of gestation". It is true that although induction of labor is familiar with obstetricians, the procedure is still raising concern from patients' side. Even in the United States where patients consulting has been routinely applied, the rate of patients refuse to be induced at 39th week of gestation is about 50%. Review from Cochrane library also suggested that "Offering women tailored counselling may help them make an informed choice between induction of labor for pregnancies" . In some countries where the National Guidelines still recommends induction of labor should be considered after 41 weeks of gestation and pregnancy related decisions are driven by many identical factors such as: knowledge, traditional or cultural ones, the patients' perspective on induction of labor before 40 weeks of gestation is a challenge. Thus, the patients' understanding of the elective induction of labor and factors contribute to decision-making process towards induction of labor should be investigated in order not only to develop appropriate induction policies for the future but also scientific studies/randomized clinical trials to come.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥ 18
* Singleton pregnancy (twin gestation reduced to singleton, either spontaneously or therapeutically, is not eligible unless the reduction occurred before 14 weeks project gestational age)
* Gestational age at 36+0 weeks to 36+6 week
* Cephalic presentation
* No contraindications to vaginal delivery

Exclusion Criteria:

1. Previous C-section
2. Maternal medical illness associated with increased risk of adverse pregnancy outcome (any diabetes mellitus, any hypertensive disorders, cardiac diseases, renal insufficiency, systemic lupus erythematosus, mental disorders, HIV positive, use of heparin or low-molecular weight heparin during the current pregnancy etc.)
3. Abnormal placenta: Active vaginal bleeding greater than bloody show or placenta previa, accreta or vasa previa
4. Abnormal amniotic fluid volume:

   Oligohydramnios (MVP < 2cm) Polyhydramnios (MVP > 10cm)
5. Abnormal fetus Fetal demise or known major fetal anomalies Fetal growth restriction (FGR) (EFW < 3% or < 10% and abnormal Doppler) Non-reassuring fetal status (no fetal movements, abnormal fetal heart rate at auscultation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Low risk pregnant women with a gestational age at 36th week and 39th weeks
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients accept to undergo elective induction of labor at 39th gestational week | It is planned to fill the questionnaire in 30 minutes at 39th gestational week
  Number of patients who are willing to undergo elective Induction of labor without maternal of fetal indication at 39th gestational week

SECONDARY OUTCOMES:
Participants knowledge | It is planned to fill the questionnaire in 30 minutes at 36th gestational week
  Description of knowledge and opinions of participants towards induction of labor The knowledge about induction of labor, consisted of 13 multiple choice questions including different methods, indications, contraindications, maternal and fetal benefits/ risks of induction of labor.
Participants opinions | It is planned to fill the questionnaire in 30 minutes at 36th gestational week
  Opinion about the needs for induction of labor, consisted of 12 questions including different reasons for labor induction. Participants choose the level of agreement (strongly disagree; disagree; support; strongly support) for each questions.
Reasons to choose or refuse elective induction of labor at 36th gestational week | It is planned to fill the questionnaire in 30 minutes at 36th gestational week
  Reasons why participants choose or refuse elective induction of labor: a checklist (yes/no) of 14 reasons and an open-end question
Reason why participants change initial decision about elective induction of labor | It is planned to fill the questionnaire in 30 minutes at 39th gestational week
  Reason why participants change decision about elective induction of labor: a checklist (yes/no) of 14 reasons and an open-end question
Factors that may affect participants' decision | It is planned to fill the questionnaire in 30 minutes at 36th gestational week
  Factors that may affect participants' decision towards elective induction of labor: multiple choice questions regarding the age, ethnic group, education background, profession, financial ability, residential and cohabitation arrangement, healthcare preferences of participants

CONTACTS AND LOCATIONS:
Overall Officials: Anh Nguyen Duy, PhD. MD, Study Director — Hanoi Obstetric and Gynecology Hospital; Ha Nguyen Thi Thu, PhD. MD, Principal Investigator — Hanoi Obstetric and Gynecology Hospital; Minh Chau Ngoc, MD, Principal Investigator — Mỹ Đức Hospital; Ben W Mol, PhD. MD, Study Chair — Monash University
Locations (1):
- Hanoi Obstetrics and Gynecology Hospital, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Result] Chen HY, Grobman WA, Blackwell SC, Chauhan SP. Neonatal and Maternal Adverse Outcomes Among Low-Risk Parous Women at 39-41 Weeks of Gestation. Obstet Gynecol. 2019 Aug;134(2):288-294. doi: 10.1097/AOG.0000000000003372. PMID 31306312
- [Result] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Result] Gallagher PJ, Liveright E, Mercier RJ. Patients' perspectives regarding induction of labor in the absence of maternal and fetal indications: are our patients ready for the ARRIVE trial? Am J Obstet Gynecol MFM. 2020 May;2(2):100086. doi: 10.1016/j.ajogmf.2020.100086. Epub 2020 Jan 12. PMID 33345957
- [Result] Middleton P, Shepherd E, Morris J, Crowther CA, Gomersall JC. Induction of labour at or beyond 37 weeks' gestation. Cochrane Database Syst Rev. 2020 Jul 15;7(7):CD004945. doi: 10.1002/14651858.CD004945.pub5. PMID 32666584